CLINICAL TRIAL: NCT04509700
Title: A Phase 2, Open-Label, Multicenter, Rollover Study to Provide Continued Treatment for Participants With B-Cell Malignancies Previously Enrolled in Studies of Parsaclisib (INCB050465)
Brief Title: Rollover Study to Provide Continued Treatment for Participants With B-Cell Malignancies Previously Enrolled in Studies of Parsaclisib (INCB050465)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 50465-801; 2022-501687-18-00 (Registry Identifier: EU CT Number); 2019-004948-30 (EudraCT Number)
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: B-Cell Malignancies
Keywords: non-Hodgkin lymphoma; phosphatidylinositol 3-kinase; myeloproliferative neoplasm
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Myeloproliferative Disorders | interventions — parsaclisib; itacitinib; ruxolitinib; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- parsaclisib (Experimental): Participants will continue on the same dose (1,2.5,5 OR 20 mg) and schedule of parsaclisib as that provided in the parent Protocol at the time of the rollover.
  Interventions: Drug: Parsaclisib
- parsaclicib + itacitinib (Experimental): Participants will continue on the same dose (1,2.5,5 OR 20 mg) and schedule of parsaclisib and 100 mg of itacitinib as that provided in the parent Protocol at the time of the rollover.
  Interventions: Drug: parsaclisib + itacitinib
- parsaclisib + ruxolitinib (Experimental): Participants will continue on the same dose (1,2.5,5 OR 20 mg) and schedule of parsaclisib and the same dose of ruxolitinib that was provided in the parent Protocol at the time of the rollover.
  Interventions: Drug: parsaclisib + ruxolitinib
- parsaclisib + ibrutinib (Experimental): Participants will continue on the same dose (1,2.5,5 OR 20 mg) and schedule of parsaclisib and 140 mg of ibrutinib as that provided in the parent Protocol at the time of the rollover.
  Interventions: Drug: parsaclisib + ibrutinib

INTERVENTIONS:
Drug: Parsaclisib — Participants will continue on the same dose (1,2.5,5 OR 20 mg) and schedule of parsaclisib as that provided in the parent Protocol at the time of the rollover.
  Other Names: INCB050465
  Arms: parsaclisib
Drug: parsaclisib + itacitinib — Participants will continue on the same dose (1,2.5,5 OR 20 mg) and schedule of parsaclisib and 100 mg of itacitinib as that provided in the parent Protocol at the time of the rollover.
  Other Names: INCB050465; INCB39110
  Arms: parsaclicib + itacitinib
Drug: parsaclisib + ruxolitinib — Participants will continue on the same dose (1,2.5,5 OR 20 mg) and schedule of parsaclisib and the same dose of ruxolitinib that was provided in the parent Protocol at the time of the rollover.
  Other Names: INCB050465; INCB018424
  Arms: parsaclisib + ruxolitinib
Drug: parsaclisib + ibrutinib — Participants will continue on the same dose (1,2.5,5 OR 20 mg) and schedule of parsaclisib and 140 mg of ibrutinib as that provided in the parent Protocol at the time of the rollover.
  Other Names: INCB050465
  Arms: parsaclisib + ibrutinib

SUMMARY:
This is a Phase 2, multicenter, open-label study to provide continued supply of parsaclisib as monotherapy or in combination therapy with itacitinib, ruxolitinib, or ibrutinib to participants from Incyte-sponsored studies of parsaclisib.

DETAILED DESCRIPTION:
The purpose of this study is to provide continued use of parsaclisib as monotherapy or in combination with itacitinib, ruxolitinib, or ibrutinib to participants who are currently enrolled in an Incyte-sponsored study and receiving the same treatment, who have at least stable disease, who are obtaining clinical benefit (in the opinion of the investigator) on the current study treatment, as defined by the parent Protocol, and who are unable to access parsaclisib as monotherapy or in combination with itacitinib, ruxolitinib, or ibrutinib outside a clinical study. Participants will continue on the same dose and schedule as the ones being administered in the Incyte-sponsored parent Protocol at the time of the rollover. The study will collect and assess safety information with regards to AEs.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled and receiving treatment in an Incyte-sponsored clinical study of parsaclisib.
* Currently tolerating treatment in the parent Protocol.
* Currently receiving clinical benefit from treatment with parsaclisib as monotherapy or in combination therapy with Itacitinib, ruxolitinib, or ibrutinib as determined by the investigator.
* Has at least stable disease, as determined by the investigator.
* Has demonstrated compliance, as assessed by the investigator, with the parent Protocol requirements.
* Willingness and ability to comply with scheduled visits, treatment plans, including PJP prophylaxis, and any other study procedures indicated in this Protocol.
* Willingness to avoid pregnancy or fathering children
* Ability to comprehend and willingness to sign an ICF

Exclusion Criteria:

* Has been permanently discontinued from study treatment in the parent Protocol for any reason.
* Able to access parsaclisib as monotherapy or in combination with itacitinib, ruxolitinib, or ibrutinib therapy outside a clinical study.
* Participants with an uncontrolled intercurrent illness or any concurrent condition that, in the investigator's opinion, would jeopardize the safety of the participant or compliance with the Protocol.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through study completion, an average of 5 years
  Number of participants with treatment-related AEs

CONTACTS AND LOCATIONS:
Locations (104):
- United States (26):
  - Uab Comprehensive Cancer Center, Birmingham, Alabama
  - University of Alabama At Birmingham, Birmingham, Alabama
  - Mayo Clinic Rochester, Phoenix, Arizona
  - University of Arizona Cancer Center-Out Pt., Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - California Cancer Associates For Research and Excellence, Fresno, California
  - Innovative Clinical Research Institute, Long Beach, California
  - Rocky Mountain Cancer Center, Aurora, Colorado
  - Rush University Medical Center-Consultants in Hematology, Chicago, Illinois
  - University of Kansas Hospital Authority, Westwood, Kansas
  - Rcca Md, Llc, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Hattiesburg Clinic Hematology, Hattiesburg, Mississippi
  - Saint Luke'S Hospital of Kansas City, Kansas City, Missouri
  - Hca Midwest Health-Research Medical Center, Kansas City, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Knight Cancer Institute At Oregon Health and Science University, Portland, Oregon
  - Baylor Scott White Univeristy Medical Center, Dallas, Texas
  - University of Washington-Seattle Cancer Care Alliance, Seattle, Washington
- Medical University of Vienna, Vienna, Austria
- Belgium (4):
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent (Uz Gent), Ghent
  - Az Groeninge, Kortrijk
  - Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven
- Czechia (4):
  - University Hospital Hradec Kralove, Hradec Králové
  - Univerzita Karlova V Praze 1. Lekarska Fakulta, Prague
  - Fakultni Nemocnice V Motole, Prague
  - University Hospital Kralovkse Vinohrady, Prague
- Denmark (3):
  - Aarhus University Hospital, Århus N
  - Rigshospitalet, Copenhagen
  - Sjaellands Universitetshospital, Roskilde
- France (6):
  - Chru de Brest Hospital Morvan, Brest
  - Centre Antoine Laccassagne, Nice
  - Ap-Hp Groupe Hospitalier Saint-Louis Lariboisiere Fernand-Widal Site Saint Louis (Paris), Paris
  - Hospital Universitaire Pitie-Salpetriere, Paris
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
  - Chru Hopitaux de Tours Hospital Bretonneau, Tours
- Petz Aladar County Teaching Hospital, Győr, Hungary
- Israel (3):
  - Hadassah Hebrew University Medical Center Ein Karem Hadassah, Jerusalem
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky
- Italy (13):
  - University of Bologna Institute of Haematology L E A Seragnoli, Bologna
  - Lstituto Di Ematologia Lorenzo Ea.Seragnoli Universita Degli Studi Di Bologna - Policlinico S. Or, Bologna
  - Azienda Ospedaliero-Universitaria Careggi (Aouc), Florence
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori, Meldola (FC)
  - Fondazione Irccs Ca Granda Ospedale Maggiore, Milan
  - Comitato Etico Fondazione Irccs Istituto Nazionale Dei Tumori Milano, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Universita Di Napoli Federico Ii, Naples
  - Azienda Ospedaliero Universitaria Maggiore Della Carita Di Novara, Novara
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - Azienda Ospedaliero Universitaria Pisana - Ospedale S. Chiara, Pisa
  - Ospedale Santa Maria Delle Croci, Ravenna
  - Ospedale Sant. Eugenio, Roma
- Japan (19):
  - Juntendo University Hospital, Bunkyō City
  - National Cancer Center Hospital, Chūō
  - Kansai Medical University Hospital, Hirakata
  - Tokai University Hospital, Isehara
  - Irb of Kobe City Medical Center General Hospital, Kobe
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Nho Matsumoto Medical Center, Matsumoto-shi
  - Miyagi Cancer Center, Miyagi
  - Jrc Aichi Medical Center Nagoya Daini Hospital, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Osaka Metropolitan University Hospital, Osaka
  - Hokuyukai Sapporo Hokuyu Hospital, Sapporo
  - National Hospital Org. Hokkaido Cancer Center, Sapporo
  - Tohoku University Hospital, Sendai
  - Tokyo Medical University Hospital, Shinjuku
  - Tenri Hospital, Tenri
  - Nippon Medical School Hospital, Tokyo
  - Yokohama Municipal Citizens Hospital, Yokohama
  - University of Fukui Hospital, Yoshida-gun
- Haukeland University Hospital, Bergen, Norway
- Poland (4):
  - Sp Zoz Szpital Uniwersytecki, Kracow
  - Wwcoit Im. M. Kopernika W Lodzi, Lodz
  - Szpital Specjalistyczny Im. Jedrzeja Sniadeckiego W Nowym Saczu, Nowy Sącz
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Wroclaw
- The Catholic University of Korea Seoul St. Mary'S Hospital, Seoul, South Korea
- Spain (14):
  - Hospital General Unviersitario de Alicante, Alicante
  - Germans Trias I Pujol, Badalona
  - Hospital Del Mar, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Start Madrid - Ciocc, Boadilla del Monte
  - Institut Catala Doncologia - Hospital Duran I Reynals, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Fundacin Jimnez Daz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Hm Sanchinarro, Madrid
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
- Karolinska University Hospital Solna, Stockholm, Sweden
- Turkey (Türkiye) (2):
  - Istanbul Medipol Universitesi Ibagcilar Medipol Mega Universitesi Hastanesi, Istanbul
  - Ege University Hospital, Izmir
- Birmingham Heartlands Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: Rollover Study to Provide Continued Treatment for Participants With B-Cell Malignancies Previously Enrolled in Studies of Parsaclisib (INCB050465) — https://incyteclinicaltrials.com/studies/incb-50465-801